CLINICAL TRIAL: NCT06480773
Title: Kaposi Sarcoma Chemotherapy and Research (KS-CARE): Clinical and Molecular Determinants of HIV-associated Kaposi Sarcoma Progression Under Local Standard-of-care Therapy in Malawi and South Africa
Brief Title: Kaposi Sarcoma Chemotherapy and Research (KS-CARE)
Acronym: KS-CARE
Status: Active, not recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: KS-CARE; U54CA254564 (NIH)
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Kaposi Sarcoma; HIV
Keywords: Paclitaxel; Bleomycin; Vincristine; anti- retroviral
MeSH Terms: conditions — Sarcoma, Kaposi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HIV-associated Kaposi Sarcoma: Patients receive standard-of-care chemotherapy.
  Interventions: Drug: standard of care chemotherapy

INTERVENTIONS:
Drug: standard of care chemotherapy — intravenous Paclitaxel or the combination of Bleomycin and Vincristine.

SUMMARY:
This prospective, nonrandomized, open-label, single-arm, cohort study examines the effects of chemotherapy provided under local standard of care in patients with pathologically confirmed HIV-associated Kaposi Sarcoma (HIV-KS). Previous HIV-KS studies demonstrated significant variability in clinical outcomes based on differences in gender or baseline KSHV DNA levels in patients with HIV-KS.

Patients will receive chemotherapy according to local site treatment guidelines and standard of care. Chemotherapy regimen for two treatments that are used locally based on physician's choice namely intravenous (IV) Paclitaxel (PTX) or the combination of Bleomycin and Vincristine (BV). In addition, all histologically proven HIV-KS could be enrolled, irrespective of their prior length of combination anti-retroviral treatment (cART). This enrolment strategy will reflect a more realistic picture of HIV-KS management.

This study result could trigger treatment alteration of HIV-KS. The treatment approaches to HIV-KS can be individualized if clinically relevant subsets and novel prognostic markers are defined. In that case, newer and potentially more expensive agents can be selectively applied to those patients most likely to benefit, especially if prolonged treatment is needed.

ELIGIBILITY:
Inclusion Criteria:

Participants meeting all the inclusion criteria listed below will be eligible for screening.

* Histologically confirmed T1 KS presenting to TBH combined Kaposi Sarcoma clinic with or without visceral disease. no evidence of improvement in human immunodeficiency virus (HIV)-associated Kaposi Sarcoma (HIV-KS) in the 4 weeks immediately prior; and a clinical indication for systemic chemotherapy treatment
* Known HIV-1 infection status, as documented by any nationally approved, licensed HIV rapid test and confirmed at any time point prior by the local standard of care assay.
* On ART or not on ART.
* Age ≥18 years.
* Participants able to understand and provide written informed consent in English, Afrikaans, or isiXhosa.

Exclusion Criteria:

Failure to meet the inclusion criteria listed above.

* Specifically, pregnancy and breastfeeding are not exclusion criteria given the observational nature of the study with diagnostic and treatment interventions administered according to local standards of care.
* Specifically, the absence of skin lesions is not an exclusion criterion if recorded evidence of
* visceral or nodal disease is present in the form of a radiology or endoscopy report.
* Participants who have had prior chemotherapy or radiotherapy for human immunodeficiency virus (HIV)-associated Kaposi Sarcoma.
* Specifically, patients who have had prior cART will not be excluded.
* Participants who are receiving any other investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with human immunodeficiency virus (HIV)-associated Kaposi Sarcoma (HIV-KS) receiving treatment at Study Site
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to 48 weeks
  PFS will be defined as first chemotherapy day until disease progression. Mucocutaneous and visceral Human immunodeficiency virus (HIV)-associated Kaposi Sarcoma (HIV-KS) response will be assessed separately according to protocol-defined definitions. Mucocutaneous Progressive disease (mcPD) is defined as any increase or progression in the size, type and/or number of skin and/or mucosal lesions if present at baseline or new lesion. Visceral Progressive disease (vPD) is defined as any increase in symptoms related to visceral HIV-KS if present at baseline or a new manifestation of symptoms related to visceral HIV-KS, not present at baseline, or radiological or endoscopic evidence of visceral KS, not present at baseline. Notably, lymphoedema and nodal disease will not be part of the formal response assessment for CR, PR, and SD response criteria should have been maintained for at least 4 weeks. For PD response criteria can have been present for at least 1 week.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) - 96 weeks | Up to 96 weeks
  PFS will be defined as the time from chemotherapy treatment initiation until disease progression. Mucocutaneous and visceral Human immunodeficiency virus (HIV)-associated Kaposi Sarcoma (HIV-KS) response will be assessed separately according to protocol-defined definitions. Mucocutaneous Progressive disease (mcPD) is defined as any increase or progression in the size, type and/or number of skin and/or mucosal lesions if present at baseline or new lesion. Visceral Progressive disease (vPD) is defined as any increase in symptoms related to visceral HIV-KS if present at baseline or a new manifestation of symptoms related to visceral HIV-KS, not present at baseline, or radiological or endoscopic evidence of visceral KS, not present at baseline. Notably, lymphoedema and nodal disease will not be part of the formal response assessment for CR, PR, and SD response criteria should have been maintained for at least 4 weeks. For PD response criteria can have been present for at least 1 week.
Response rates (ORR) | Up to 4 weeks
  Response rate will be assessed by Mucocutaneous and visceral Human immunodeficiency virus (HIV)-associated Kaposi Sarcoma (HIV-KS) separately according to protocol-defined definitions. ORR = Partial response (PR) or complete response (CR). Muco-Cutaneous Complete response (mcCR) is defined as the regression of all skin and/or mucosal lesions to hyperpigmented patches or macules if present at baseline. Muco-Cutaneous Partial response (mcPR) is defined as any reduction in the size, type and/or number of skin and/or mucosal lesions if present at baseline and no new manifestation of skin and/or mucosal lesions, not present at baseline. Visceral Complete response (vCR) is defined as the absence of symptomatic visceral KS if present at baseline. Visceral Partial response (vPR) is defined as any reduction in symptoms related to visceral HIV-KS if present at baseline and no new manifestation of symptoms related to visceral HIV-KS, not present at baseline.
Overall Survival (OS) | Up to 96 weeks
  OS will be defined as the time from chemotherapy treatment initiation until death.
Health-related Quality of Life (HR-QOL) | Baseline, 4 weeks, 48 weeks, 76 weeks, 96 weeks
  HR-QOL will be measured by validated Human immunodeficiency virus (HIV)-associated Kaposi Sarcoma (HIV-KS) Functional Assessment of HIV (FAHI) Quality of Life instrument with 3 supplemental questions addressing pain, swelling, and satisfaction with physical appearance (FAHI+KS) as developed by the National Institutes of Health, will be used to collect quality of life (QOL) data in 5 categories: physical well-being, emotional well-being, functional and global well-being, social well-being, and cognitive functioning. Items are rated by patients on a Likert scale from 0 to 4. Higher scores represent worse QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Dittmer, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (2):
- UNC Project, Kamuzu Central Hospital, Lilongwe, Malawi
- Stellenbosch University and Tygerberg Hospital, Cape Town, Stellenbosch, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials